CLINICAL TRIAL: NCT05321966
Title: The Effect of Video Training on Symptom Burden, Comfort Level and Quality of Life in Patients Undergoing Hemodialysis Treatment
Brief Title: The Effect of Video Training on Symptom Burden Patients Undergoing Hemodialysis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halise Taskın Duman (Other)
Responsible Party: Sponsor-Investigator, Halise Taskın Duman, The Effect of Video Training on Symptom Burden, Comfort Level and Quality of Life in Patients Undergoing Hemodialysis Treatment, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FethiyeHSF
Record Dates: First submitted 2022-03-25; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Symptom Cluster; Quality of Life; Conformity, Social
Keywords: Hemodialysis; Visual Education; Symptom Burden; Patient Comfort; Quality of Life
MeSH Terms: conditions — Syndrome; Social Conformity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual Education Group (Experimental): The intervention group watched three episodes of a training video a week for 12 weeks. Each session started 90 minutes after the HD treatment
  Interventions: Other: Visual video education
- no intervention (No Intervention): No intervention was made to the individuals in the control group.

INTERVENTIONS:
Other: Visual video education — The intervention group watched three episodes of a training video a week for 12 weeks. Each session started 90 minutes after the HD treatment
  Arms: Visual Education Group

SUMMARY:
Purpose: This study aimed to examine the impacts of video training support on the symptom burden, comfort level and quality of life (QoL) of the patients undergoing hemodialysis (HD) treatment. Methods: The current study adopted a randomized controlled quasi-experimental research design to investigate the implications of video training support on the symptom burden, comfort level and QoL of 48 participant patients, 22 of whom were in control and 26 were in intervention group, at Mugla Fethiye State Hospital Hemodialysis Center and a private hemodialysis center between April 2021 and July 2021. Data collection was conducted through Dialysis Symptom Index (DSI), Patient Information Form, QoL Scale Short Form (SF 36), and Hemodialysis Comfort Scale (HDCS) Version II. The data was collected four times, in week 0 (1st measurement), 4th week (2nd measurement), 8th week (3rd measurement), and 12th week (4th measurement). The intervention group watched three episodes of a training video a week for 12 weeks. Each session started 90 minutes after the HD treatment. The control group was shown the training video at the end of the research. Necessary ethics committee, institutional permissions and written consents of the participant patients were obtained prior to the study.

DETAILED DESCRIPTION:
The purpose of hemodialysis treatment; to remove metabolic wastes from the blood, to reduce symptoms and complications in patients, and to increase life expectancy and quality. During HD treatment, many comorbidities, complications and symptoms may occur in patients. Alvarez et al. (2020) found diabetes and hypertension as comorbid diseases in the majority of the patients, and the most common symptoms were found to be fatigue, cramps, hypotension, headache, itching, difficulty concentrating, and dizziness.

In order to increase the success of hemodialysis treatment, the patient should make a lifestyle change, comply with the treatment and his family should support the patient. Compliance with treatment is ensured by the cooperation of the healthcare team with the patient and their relatives. As treatment compliance increases, symptom burden, complication and mortality rates decrease. For this, patients should be provided with planned trainings that are repeated at the beginning of HD treatment and at regular intervals thereafter.

The purpose of patient education; To create a healthy behavioral change in patients, to enable healthcare professionals to establish a more efficient relationship with the patient and his family, to increase the quality of life of the patient and his family, to increase the comfort of life, compliance with treatment, to reduce morbidity and mortality, and to reduce the cost of health expenses. In our country, there is no standard educational content and training calendar in HD units. Most of the lives of HD patients are spent in dialysis units. The majority of the patients spend their time in the dialysis unit for an average of four hours a day, three days a week, depending on the machine. For this reason, it is important for patients to give the training to be given during the dialysis sessions.

The research was carried out as a randomized controlled quasi-experimental study with the aim of examining the effect of video education support on patients who were treated with HD on symptom burden, comfort level and quality of life. The research was carried out in Muğla Fethiye State Hospital Hemodialysis Center and Private Fethiye Can Dialysis Center between April 2021 and July 2021. The universe of the research; Patients who received treatment at Fethiye State Hospital Hemodialysis Center and Private Fethiye Can Dialysis Center were formed. The number of patients in Fethiye State Hospital Hemodialysis Center is 44, the number of patients in Private Can Dialysis Center is 137, and a total of 181 patients receive hemodialysis treatment in two centers.

Sample of the Research; The sample size of the study was 0.25 effect size, 0.05 error level, 95% confidence interval and 95% power of 4 measurements in both groups, 18 interventions and 18 control groups, in order to be able to analyze the variance in repeated measurements within the factors in the study by using the G power 3.1.5 software program. It has been calculated that a total of 36 participants are needed.

Simple random sampling method was used in the randomization of the study. The individuals in the study were divided into clusters according to the session days. After clustering, a simple random draw (by flipping a coin) was drawn to determine which cluster would be in the intervention group and which cluster would be in the control group. The advantage of this sampling method is that it is simple and easy to implement.

Preparation of Training Video Content The topics to be included in the content of the training video were determined according to the educational needs of the patients by making a literature review (TND reports, KDIGO guidelines, research articles).

Education subject titles; Fistula description, dry weight description, fluid intake and weight control, diet, medication, skin care, oral care, exercises, infections, Sexual life

Data Collection An episode of video was watched by the intervention group, 90 minutes after the start of HD, in each session three days a week for 12 weeks. In the weekly training plan of the initiative group; The weekly training process was completed by watching a total of 3 training videos per week. No intervention was made in the control group.

The patients in the intervention group were provided with external memory and individual headphones for video monitoring. External memories were not given to the patients, they were only used by the researcher during the study.

The data were collected by the principal investigator by means of a face-to-face interview and a question-answer questionnaire method, after obtaining the written consent of the patients. At the beginning of the study, the patients in the control and intervention groups were given the Patient Identification Form, Dialysis Symptom Index, Hemodialysis Comfort Scale Version-II, Quality of Life Scale Short Form (SF 36) has been applied. At the end of the fourth, eighth and twelfth weeks, Dialysis Symptom Index, Hemodialysis Comfort Scale-Version II, Quality of Life Scale Short Form (SF 36) were applied to both groups. Data collection time lasted an average of 15-20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* Patients who have been treated for HD for 12 months or more

Exclusion Criteria:

* younger than 18,
* Initiation of HD treatment is less than 12 months,
* Vacation in HD center is within the scope of dialysis and less than 12 weeks that will come,
* Known hearing or vision problems,
* Patients with cognitive impairment,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
The change in symptom burden in hemordialysis patients | Once a month/3 times
  The dialysis-related symptoms of the patients were evaluated with the Dialysis Symptom Index. This scale is used by individuals in the last seven days. He questions his symptoms. The scale consists of 30 questions in 5-point Likert type. An increase in the scale score is symptom indicates an increased load.
The change in comfort level in hemodialysis patients | Once a month/3 times
  Hemodialysis Comfort Scale Version II scale is a 5-point Likert type scale consisting of 26 items and six sub-dimensions. As the scale score increases, comfort increases, while as the score decreases, comfort decreases. The scale score range is min-max= 26-130 points. The scale consists of 6 dimensions in total. These dimensions are physical relaxation, physical relaxation, psychospiritual relaxation, psychospiritual empowerment, environmental empowerment, sociocultural relaxation.
The change in quality of life in hemodialysis patients | Once a month/3 times
  The impairment in the patients' quality of life was evaluated with the Short Form of the Quality of Life Scale (SF 36). The scale consists of 36 questions and the last four weeks of the individuals are questioned. The scale consists of eight sub-dimensions. These dimensions are; physical function, physical role difficulty, emotional role difficulty, energy/vitality/vitality, mental health, social functionality, pain, general health perception. Each of the sub-dimensions is evaluated separately. On the scale, "0" indicates poor health, "100" indicates good health.

CONTACTS AND LOCATIONS:
Overall Officials: Halise Taskin Duman, Phd, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Mugla Sitki Kocman University, Muğla, Fethiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No